CLINICAL TRIAL: NCT01980849
Title: Phase Ⅲ Study of Prophylaxis of Venous Thromboembolism in Advanced Lung Cancer by Nadroparin
Brief Title: Prophylaxis of Venous Thromboembolism in Advanced Lung Cancer
Acronym: LCAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengqing Li (Other)
Responsible Party: Sponsor-Investigator, Shengqing Li, Consultant, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LCAN-20131105
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Lung Cancer
Keywords: Nadroparin; venous thromboembolism prophylaxis
MeSH Terms: conditions — Lung Neoplasms | interventions — Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long term prophylaxis (Experimental): Nadroparin, 0.4mL, subcutaneously, qid, given by long-term
  Interventions: Drug: Nadroparin, long term
- Short-term prophylaxis (Active Comparator): Nadroparin, 0.4mL, subcutaneously, qid, given during hospitalization
  Interventions: Drug: Nadroparin: short-term

INTERVENTIONS:
Drug: Nadroparin, long term
  Arms: Long term prophylaxis
Drug: Nadroparin: short-term
  Arms: Short-term prophylaxis

SUMMARY:
To compare the efficacy and safety of prophylaxis of venous thromboembolism by Nadroparin during hospitalization to long-term usage in patients with advanced lung cancer treated by chemotherapy and/or radiotherapy.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized and controlled study. Advanced lung cancer patients without venous thromboembolism(VTE) are included. The selected patients were randomized into A and B groups. Group A: Nadroparin given during hospitalization, 0.4mL, subcutaneously, qid; Group B: Nadroparin given by long-term, 0.4mL, subcutaneously, qid. The incidence of VTE , the risks of bleeding and overall survival in two groups of patients are studied at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Stage Ⅲ B and Ⅳ non-small cell lung cancer patients and inoperable small cell lung cancer patients
* Performance status score ≤ 2
* Chest CT with measurable lesions

Exclusion Criteria:

* Examination revealed any part of venous thromboembolism
* Chemotherapy regimens containing bevacizumab or Endostar
* Severe coagulopathy
* Active bleeding within two weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism | 12 weeks

SECONDARY OUTCOMES:
Incidence of bleeding | During 6 months

OTHER OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The Department of Oncology，Southwest Hospital, Chongqing, Chongqing Municipality
  - The Department of Pulmonary and Critical Care Medicine,Southwest Hospital, Chongqing, Chongqing Municipality
  - The Department of Oncology，Ohtsubo Hospital, Chongqing, Chongqing Municipality
  - The Department of Oncology，Fuling Central Hospital, Chongqing, Chongqing Municipality
  - The Department of Oncology，Central Hospital, Xinxiang, Henan
  - The Department of Oncology，People's Hospital, Zhengzhou, Henan
  - The Department of Pulmonary and Critical Care Medicine,Cancer Hospital, Zhengzhou, Henan
  - The Department of Oncology，Henan University Affiliated Yihe Hospital, Zhengzhou, Henan
  - The Department of Oncology，Cancer Hospital, Baotou, Inner Mongolia
  - The Department of Oncology，Northern Hospital, Baotou, Inner Mongolia
  - The Department of Oncology，Inner Mongolia Autonomous Region Hospital, Hohhot, Inner Mongolia
  - The Department of Pulmonary and Critical Care Medicine,Medical University General Hospital cardiovascular and cerebrovascular disease hospital, Yinchuan, Ningxia
  - The Department of Pulmonary and Critical Care Medicine,Central Hospital, Baoji, Shaanxi
  - The Department of Pulmonary and Critical Care Medicine,Second People's Hospital, Xi'an, Shaanxi
  - The Department of Pulmonary and Critical Care Medicine, Second Affiliated Hospital of Jiaotong University, Xi'an, Shaanxi
  - The Department of Pulmonary and Critical Care Medicine, Tangdu Hospital, Xi'an, Shaanxi
  - The Department of Pulmonary and Critical Care Medicine, Xijing Hospital, Xi'an, Shaanxi
  - The Department of Oncology，First Affiliated Hospital of Jiaotong University, Xi'an, Shaanxi
  - The Department of Oncology，Yan'an University Hospital, Yan’an, Shaanxi
  - The Department of Oncology，Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Department of Lung oncology，Tumor Hospital, Chengdu, Sichuan
  - The Department of Oncology，People's Hospital, Chengdu, Sichuan
  - The Department of Oncology，First Affiliated Hospital of Medical University, Ürümqi, Xinjiang
  - The Department of Pulmonary and Critical Care Medicine,First Affiliated Hospital of Medical University, Ürümqi, Xinjiang